CLINICAL TRIAL: NCT02978833
Title: Ultrasound-Guided Platelet Rich Plasma Versus Whole Blood Injection for the Treatment of Gluteus Medius Tendinopathy: A Double-Blind Randomized Controlled Study
Brief Title: Platelet-rich Plasma vs. Whole Blood for Gluteus Medius Tendinopathy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow enrollment, lack of patients
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-184
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Tendinopathy; Hip Pain
Keywords: Gluteus Medius Tendinosis
MeSH Terms: conditions — Tendinopathy | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- PRP (Experimental)
  Interventions: Biological: PRP; Device: Ultrasound
- Whole Blood (Active Comparator)
  Interventions: Biological: Whole Blood

INTERVENTIONS:
Biological: PRP
  Arms: PRP
Biological: Whole Blood
  Arms: Whole Blood
Device: Ultrasound
  Arms: PRP

SUMMARY:
Gluteus medius tendinopathy, which is often referred to as Greater Trochanteric Pain Syndrome, is characterized by pain in the lateral aspect of the hip that is aggravated by side lying, stair climbing, and walking. Treatment is currently limited to lifestyle modifications, corticosteroid injections, physical therapy, and open and endoscopic surgical repair. Platelet rich plasma (PRP) injections contain important growth factors that are essential in the healing and tissue formation processes. However, the extent to which PRP is more efficacious than whole blood in tendinopathy remains unclear. In this double-blind randomized trial, patients will be allocated to receive either a PRP or whole-blood injection. Post-procedure assessments will occur at 6 weeks, 3 months, 6 months, 9 months, and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe lateral hip pain for greater than 3 months
* Symptoms are refractory to conservative treatment, including at least 8 weeks of traditional physical therapy for this condition
* Moderate to severe gluteus medius tendinosis with or without partial tear <1 cm
* Normal neurologic exam except for hip abductor weakness on the affected side

Exclusion Criteria:

* Severe (Tonnis grade >1) hip osteoarthritis with active synovitis or bone edema
* Active lumbar radiculopathy with pain, numbness or weakness in a dermatomal distribution
* No evidence of fatty atrophy, denervation, or complete tears of gluteus medius seen on MRI
* Any condition that requires anti-platelet or anti-coagulation therapy, including aspirin therapy for cardiac conditions
* Non-English speaking

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-10-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Moley, M.D., Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Platelet-rich Plasma: PRP
  Ultrasound
- Whole Blood: Whole Blood
Period: Overall Study
Arm/Group | Platelet-rich Plasma | Whole Blood
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Study terminated | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Platelet-rich Plasma | Whole Blood | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Pain
Description: The Numerical Rating Scale for Pain will be used, where 0=no pain and 10=worst pain. A higher number represents more pain.
Time Frame: Up to 1 year post-injection
Population: This study was terminated early, and data collection could not be completed. Thus, no data were analyzed.
Arm/Group | Platelet-rich Plasma | Whole Blood
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Improvement in Function
Description: The Non-Arthritic Hip Score and Veterans RAND 12-Item Health Survey will be used to assess improvement in function.
Time Frame: Up to 1 year post-injection
Population: This study was terminated early, and data collection could not be completed. Thus, no data were analyzed.
Groups:
- Platelet-rich Plasma: PRP
Arm/Group | Platelet-rich Plasma | Whole Blood
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Patient Satisfaction
Description: The 10-cm Visual Analog Scale for patient satisfaction will be used. This scale will range from "very dissatisfied" to "extremely satisfied".
Time Frame: Up to 1 year post-injection
Population: This study was terminated early, and data collection could not be completed. Thus, no data were analyzed.
Arm/Group | Platelet-rich Plasma | Whole Blood
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Quality of Movement During the Forward Step-down Test
Description: The quality of movement will be assessed on a scale of 0-4+, where 4+="good", 2-3="moderate", and 0-1="poor".
Time Frame: Up to 1 year post-injection
Population: This study was terminated early, and data collection could not be completed. Thus, no data were analyzed.
Arm/Group | Platelet-rich Plasma | Whole Blood
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Pain During Side-lying Hip Abduction
Description: Pain will be assessed using the 10-cm Visual Analog Scale, which will range from "no pain" to "worst possible pain".
Time Frame: Up to 1 year post-injection
Population: This study was terminated early, and data collection could not be completed. Thus, no data were analyzed.
Arm/Group | Platelet-rich Plasma | Whole Blood
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Pain During Forward Step-down Test
Description: Pain will be assessed using the 10-cm Visual Analog Scale, which will range from "no pain" to "worst possible pain".
Time Frame: Up to 1 year post-injection
Population: This study was terminated early, and data collection could not be completed. Thus, no data were analyzed.
Arm/Group | Platelet-rich Plasma | Whole Blood
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: This study was terminated early. Adverse event data were not collected to completion for each of the patients.
Arm/Group | Platelet-rich Plasma | Whole Blood
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT02978833/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT02978833/SAP_001.pdf